CLINICAL TRIAL: NCT02216136
Title: A Prospective Trial to Assess Tumor :Breast Ratio and Patient Satisfaction in Following Lumpectomy Versus Mastectomy With Reconstruction
Brief Title: Tumor: Breast Ratio Study
Acronym: T:B
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201404004
Record Dates: First submitted 2014-08-04; First posted 2014-08-13 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer; LCIS; DCIS
Keywords: Mastectomy; Breast Cancer; Reconstruction; Lumpectomy; Breast Conservation Therapy
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Breast Conservation Cohort: Breast Conservation group (Group A) with newly diagnosed breast cancer who decide to proceed with lumpectomy and radiation treatment.
- Mastectomy and Reconstruction Cohort: Mastectomy and Reconstruction group (Group B): This group will have mastectomy with immediate reconstruction (defined as reconstruction process starting at time of initial mastectomy surgery). They may or may not require chemotherapy and radiation depending on their cancer staging as well as multiple steps of their breast reconstruction.
- Mastectomy Only Cohort: Mastectomy Only Cohort: This group will have mastectomy without reconstruction. They may or may not require chemotherapy and radiation.

SUMMARY:
This is an observational study of 3 arms: breast conservation therapy, mastectomy and reconstruction, and mastectomy only.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be scheduled to undergo breast conservation therapy (BCT), mastectomy or mastectomy with immediate reconstruction (defined as initiating the reconstructive process at time of mastectomy) for ductal carcinoma in situ (DCIS), lobular carcinoma in situ (LCIS), and early stage breast cancer (Clinical Stages IA-IIB). Stage IIB tumors are 2-5 cm with micrometastases 0.2 to 2.0 cm in lymph nodes; or 2-5 cm tumor with 1-3 positive axillary or internal mammary lymph nodes, or >5 cm with no lymph node involvement. Clinical staging, based on imaging and physical exam will be used for enrollment. Patients that are upstaged due to unexpected findings at the time of surgery/assessment of surgical pathology will be excluded at that time. For staging reference please see http://www.cancer.gov/cancertopics/pdq/treatment/breast/patient/page2#keypoint13
* If multifocal/multicentric disease of the ipsilateral breast is encountered and patients are still deemed eligible for BCT or mastectomy per standard of care, then the tumor area will be calculated as the total volumes of the identified foci.
* Patient must be between 18-72 years old
* Patient must be able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Cognitive impairment
* History of radiation to the chest wall or breasts
* Patients unable to undergo MRI due to metallic implant or claustrophobia
* Patients that are pregnant since breast MRI is contraindicated
* History of previous breast surgery other than primary cosmetic augmentation or breast reduction
* Identification of a concurrent or synchronous contralateral cancer during the enrollment period
* Any patient that would not have been considered for BCT or reconstruction
* BCT patients planning to proceed with reconstruction during their study participation timeline

Ages: 18 Years to 72 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females ages 18 - 72 years of age scheduled to undergo breast conservation therapy (BCT), mastectomy or mastectomy with immediate reconstruction for ductal carcinoma in situ (DCIS), lobular carcinoma in situ (LCIS), and early stage breast cancer (Clinical Stages IA-IIB).
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence M. Myckatyn, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Dolen U, Thornton M, Tenenbaum MM, Aripoli A, Patel A, Cyr AE, Yan Y, Appleton CM, Margenthaler JA, Myckatyn TM. A prospective cohort study to analyze the interaction of tumor-to-breast volume in breast conservation therapy versus mastectomy with reconstruction. Breast Cancer Res Treat. 2020 Jun;181(3):611-621. doi: 10.1007/s10549-020-05639-w. Epub 2020 Apr 30. PMID 32350679
- See also: This website allows for direct access to the West County Plastic Surgeons' web site. — http://westcountyplasticsurgeons.wustl.edu/
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mastectomy Only cohort was unable to enroll participants due to: participants who chose mastectomy with no reconstruction almost never had an MRI and MRI was a critical inclusion criteria; most of the participants who were approached were older and refused participation; issue with finding and tracking participants who refused reconstruction
Groups:
- Breast Conservation Cohort: Breast Conservation group with newly diagnosed breast cancer who decide to proceed with lumpectomy and radiation treatment.
- Mastectomy and Reconstruction Cohort: Mastectomy and Reconstruction group: This group will have mastectomy with immediate reconstruction (defined as reconstruction process starting at time of initial mastectomy surgery). They may or may not require chemotherapy and radiation depending on their cancer staging as well as multiple steps of their breast reconstruction.
Period: Overall Study
Arm/Group | Breast Conservation Cohort | Mastectomy and Reconstruction Cohort | Mastectomy Only Cohort
Started | 72 | 90 | 0
Completed | 72 | 90 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Mastectomy Only cohort was unable to enroll participants due to: participants who chose mastectomy with no reconstruction almost never had an MRI and MRI was a critical inclusion criteria; most of the participants who were approached were older and refused participation; issue with finding and tracking participants who refused reconstruction
Groups:
- Total: Total of all reporting groups
Arm/Group | Breast Conservation Cohort | Mastectomy and Reconstruction Cohort | Mastectomy Only Cohort | Total
Number analyzed (Participants) | 72 | 90 | 0 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (8.8) | 54.7 (10.5) |  | 54.6 (25.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 90 |  | 162
  Male | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 |  | 9
  Asian | 3 | 3 |  | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 4 | 4 |  | 8
  White | 58 | 79 |  | 137
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 2 | 0 |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 72 | 90 |  | 162

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life as Measured by the Breast Q
Description: The Breast Q is a comprehensive and specific quality of life instrument that allows for patient self-assessment prior to and following breast surgery. Comprised of quality of life and satisfaction domains, and generates domain-specific Q-scores (0-100) constructed using Rasch analysis. The higher the score, the more satisfied the participant was.
  -Collected preoperatively (no more than 3 months prior to surgery) and postoperatively (approximately 6 months after conclusion of radiotherapy in the Breast Conservation Cohort and >=3 months after the final balancing reconstructive intervention in the Mastectomy and Reconstruction Cohort.
Time Frame: Compare preoperative values with postoperative values (up to 4 years)
Population: -Mastectomy Only cohort was unable to enroll participants due to: participants who chose mastectomy with no reconstruction almost never had an MRI and MRI was a critical inclusion criteria; most of the participants who were approached were older and refused participation; issue with finding and tracking participants who refused reconstruction
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breast Conservation Cohort | Mastectomy and Reconstruction Cohort | Mastectomy Only Cohort
Number analyzed (Participants) | 72 | 90 | 0
score on a scale
  Satisfaction with breasts (preop): number analyzed (Participants) | 51 | 81 | 0
  Satisfaction with breasts (preop) | 61.9 (20.4) | 57.6 (17.1) |
  Satisfaction with breasts (postop): number analyzed (Participants) | 47 | 75 | 0
  Satisfaction with breasts (postop) | 74.2 (19.8) | 64.2 (16.8) |
  Psychosocial well-being (preop): number analyzed (Participants) | 52 | 81 | 0
  Psychosocial well-being (preop) | 68.6 (16.0) | 66.8 (14.6) |
  Psychosocial well-being (postop): number analyzed (Participants) | 47 | 75 | 0
  Psychosocial well-being (postop) | 81.4 (21.7) | 72.6 (18.6) |
  Sexual well-being (preop)): number analyzed (Participants) | 51 | 80 | 0
  Sexual well-being (preop)) | 62.4 (20) | 57.5 (19.4) |
  Sexual-well being (postop): number analyzed (Participants) | 45 | 74 | 0
  Sexual-well being (postop) | 64.5 (15.8) | 54.4 (20.4) |

ADVERSE EVENTS:
Time Frame: This is an observational study as such adverse events were not collected.
Description: This is an observational study as such adverse events were not collected.
Arm/Group | Breast Conservation Cohort | Mastectomy and Reconstruction Cohort | Mastectomy Only Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT02216136/Prot_SAP_000.pdf